CLINICAL TRIAL: NCT04975490
Title: Beobachtungsstudie für Die Charakterisierung Der Pathogenese Des Akut-auf-chronischen Leberversagens
Brief Title: Characterization and Pathogenesis of ACLF
Acronym: ACLF-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Jonel Trebicka, Principal Investigator and Coordinator, Johann Wolfgang Goethe University Hospital
Other Study IDs: ACLF-Initiative
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Liver Cirrhosis; Acute-On-Chronic Liver Failure; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SAPIENT = Sepsis ACLF patients
- PROACT = Portal mediators as ACLF Targets
- ELITE = prEdictors of beneficial LIver Tx in ACFL patiEnts

SUMMARY:
This single-center prospective observational study aims at characterization of pathogenesis of ACLF. There will be three different cohorts investigated with the main endpoint mortality in these groups.

1. SAPIENT = Sepsis ACLF patients, to investigate the differences between ACLF and sepsis in cirrhosis
2. PROACT = Portal mediators as ACLF Targets, to assess portal venous biomarkers in patients receiving TIPS leading to ACLF and identify potential treatment targets
3. ELITE = prEdictors of beneficial LIver Tx in ACFL patiEnts, to assess in ACLF-patients receiving liver transplantation predictors of survival, which may improve selection of ACLF-patients for liver transplantation Secondary endpoints will be different in the three different cohorts and biological material will be collected for separate ancillary studies.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis

Exclusion Criteria:

* extrahepatic and metastatic malignancy,
* refusal for participation
* decision of attending phycisian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with liver cirrhosis and complications
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jonel Trebicka, MD, PhD, Principal Investigator — Goethe University Hospital Frankfurt
Locations (1):
- Translational Hepatology, Frankfurt am Main, Hesse, Germany